CLINICAL TRIAL: NCT03706612
Title: Shape Up! Kids Study
Status: Completed | Type: Observational
Sponsor: University of Hawaii (Other)
Collaborators: University of California, San Francisco (Other); Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: R01DK111698 (NIH)
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Identify the unique associations of body shape to body composition and bone density indices in a pediatric population that represents the variance of sex, age, BMI-Z, and ethnicity found in the US population.

Describe the precision and accuracy of optical scans to monitor change in body composition, bone density and metabolic health interventions.

Estimate the level of association of optical to common health indicators including metabolic risk factors (glucose, triglycerides, HDL-cholesterol, blood pressure, VAT, WC and strength) by gender, race, age, and BMI-Z.

Investigate holistic, high-resolution descriptors of 3D body shape as direct predictors of body composition and metabolic risk using statistical shape models and Latent Class Analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants will be included in the study if they have a self-reported ability to:

  * walk one-quarter of a mile and climb 10 steps without difficulty,
  * perform activities of daily living (ADLs) without difficulty, and
  * have no life-threatening conditions or diseases that would alter body composition from what is typical for age, sex, ethnicity, and BMI.

Exclusion Criteria:

* any internal metal artifact (e.g. pacemakers, internal fixation, arthroplasty), amputation, physical impairment or previous fracture that would alter body composition assessment
* Pregnant or breastfeeding. (All premenopausal females will be asked for a spot urine sample for pregnancy test prior to participation. Those unwilling to comply with this will not be included.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigator will recruit a stratified sample of 720 participants, approximately 360 from each site, using the following equally-weighed stratifications: sex, age (5-10, 11-14, 15-17 years), BMI-Z score (less than -2, -2 to 1, 1 to 2, and greater than 2) and ethnicity (White, Black, Mexican-American, Asian and Native Hawaiian or Other Pacific Islander).
  Within this sample, the investigator will include up to 36 participants with very low and high BMI by special recruitments from the facilities. The remainder of the participants will be recruited as a sample of convenience using local advertisements around the specified facilities.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Fat mass by DXA | 1 day
  Measure fat mass and percent fat (arms, legs, trunk, and total) using Dual energy X-ray absorptiometry (DXA) data
Lean mass by DXA | 1 day
  Measure lean mass (arms, legs, trunk, and total) using Dual energy X-ray absorptiometry (DXA) data
Bone mass by DXA | 1 day
  Measure bone mass (arms, legs, lumbar spine, and total) and Bone Mineral Density (spine and total) using Dual energy X-ray absorptiometry (DXA) data
Fat mass by MRI | 1 day
  Measure fat mass and percent fat (arms, legs, trunk, visceral, and total) using MRI data
Lean mass by MRI | 1 day
  Measure lean mass (arms, legs, trunk, and total) using MRI data
Waist to Hip ratio (WHR) from manual tape measurement | 1 day
  Manual physical anthropometry of waist and hip circumferences
Automatic 3D optical (3DO) scan measurement | 1 day
  Automated 3DO measurement generated across the body
Hand-grip strength | 1 day
  Measured by using a hand-grip dynamometer (JAMAR) as a measure of strength and physical capacity.
Isokinetic peak torque | 1 day
  Measure the peak torque value (FT-LBS) generated during isokinetic knee extension/flexion movement evaluation at 60 degrees will be assessed with the HUMAC NORM device
Isometric peak torque | 1 day
  Measure the peak torque value (FT-LBS) generated during isometric knee extension/flexion movement evaluation at 60 degrees will be assessed with the HUMAC NORM device
Fasting glucose levels | 1 day
  Measure fasting glucose levels
Fasting HbA1c levels | 1 day
  Measure fasting HbA1c levels
Fasting insulin levels | 1 day
  Measure fasting insulin levels
Fasting cholesterol levels | 1 day
  Measure fasting cholesterol levels
Fasting triglycerides levels | 1 day
  Measure fasting triglycerides levels

SECONDARY OUTCOMES:
Fat loss | 24 weeks
  Measure changes in fat mass during intervention using DXA data.
Changes in lean mass | 24 weeks
  Measure changes in lean mass (arms, legs, trunk, and total) during intervention using DXA data.
Changes in WHR | 24 weeks
  Measure changes in WHR during intervention
Changes in automatic 3DO scan measurement | 24 weeks
  Changes of automated 3DO measurements during intervention
Changes in isokinetic peak torque | 24 weeks
  Measure the change in peak torque value generated during isokinetic knee extension/flexion movement evaluation at 60 degrees will be assessed with the HUMAC NORM device pre and post intervention.
Changes in isometric peak torque | 24 weeks
  Measure the change in peak torque value generated during isometric knee extension/flexion movement evaluation at 60 degrees will be assessed with the HUMAC NORM device pre and post intervention
Total Body Water | 24 weeks
  Measure total body water (L) provided by bioelectrical impedance analysis
Phase angle | 24 weeks
  Phase angle [PhA(°) = (reactance/electrical resistance) × (180°/Π)] will be measured in degrees using bioelectrical impedance analysis.
Percent body fat | 24 weeks
  Measure percent body fat provided by bioelectrical impedance analysis.
Body circumference from 2D imaging | 24 weeks
  A conventional digital camera will be used to capture 2D images of participants in a standardized pose. Body circumference will be estimated using these images.
Systolic and Diastolic blood pressure levels will be assessed | 24 weeks
  Manually measure systolic and diastolic blood pressure levels.
Diet History Questionnaire II | 24 weeks
  The Diet History Questionnaire II estimates the participants nutrition intake by asking the participant a series of questions

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana

REFERENCES:
- [Derived] Marazzato F, McCarthy C, Field RH, Nguyen H, Nguyen T, Shepherd JA, Tinsley GM, Heymsfield SB. Advances in digital anthropometric body composition assessment: neural network algorithm prediction of appendicular lean mass. Eur J Clin Nutr. 2024 May;78(5):452-454. doi: 10.1038/s41430-023-01396-3. Epub 2023 Dec 23. PMID 38142263
- [Derived] Bennett J, Wong MC, McCarthy C, Fearnbach N, Queen K, Shepherd J, Heymsfield SB. Emergence of the adolescent obesity epidemic in the United States: five-decade visualization with humanoid avatars. Int J Obes (Lond). 2022 Sep;46(9):1587-1590. doi: 10.1038/s41366-022-01153-9. Epub 2022 May 24. PMID 35610336
- [Derived] Wong MC, Ng BK, Kennedy SF, Hwaung P, Liu EY, Kelly NN, Pagano IS, Garber AK, Chow DC, Heymsfield SB, Shepherd JA. Children and Adolescents' Anthropometrics Body Composition from 3-D Optical Surface Scans. Obesity (Silver Spring). 2019 Nov;27(11):1738-1749. doi: 10.1002/oby.22637. PMID 31689009